CLINICAL TRIAL: NCT04526717
Title: Phase 1, Open Label, Single Arm Study to Evaluate the Safety, Tolerability and Efficacy of MPT0B640 in Patients With COVID-19 Infection
Brief Title: Heat Shock Protein Inhibitor- MPT0B640 for COVID-19 Infection
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was determined not to initiate.
Sponsor: J Ints Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JO201901-02
Record Dates: First submitted 2020-07-30; First posted 2020-08-26 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Classical 3+3 design to determine MTD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MPT0B640 (Other): There is single Arm in this clinical trials.
  Interventions: Drug: MPT0B640

INTERVENTIONS:
Drug: MPT0B640 — Each dose of MPT0B640 will be administrated per Cohort. (15, 30, 60, 80, 100 mg of MPT0B640)

SUMMARY:
Indication : Treatment of Subject with COVID-19 infection Phase : Phase I Duration of Study : 12 day Sample size : at least 15 subjects Methodology : Classical 3+3 design Investigational Product : MPT0B640, 15, 30, 60, 80 and 100mg, oral suspension Study Objective

1. Primary Objective To determine the maximum tolerated dose (MTD) or maximum feasible dose (MFD) of MPT0B640
2. Secondary Objectives To evaluate the safety and tolerability of MPT0B640 during entire study period To assess the efficacy of MPT0B640 To characterize the 48 hours PK of MPT0B640

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all inclusion criteria as listed below:

1. Age ≥18 years at time of signing Informed Consent Form
2. Laboratory (quantitative Polymerase Chain Reaction, qPCR) confirmed infection with 2019-nCoV.
3. Lung involvement confirmed with chest imaging
4. Hospitalized with a SaO2/SPO2≤94% on room air or PaO2/FiO2 ratio <300mgHg
5. ≤7 days since illness onset
6. Must agree not to enroll in another study of an investigational agent prior to completion of Day 12 of study.

Exclusion Criteria:

1. Physician makes a decision that trial involvement is not in patients' best interest, or any condition that does not allow the protocol to be followed safely.
2. Severe liver disease (e.g. Child Pugh score ≥ C, AST>5 times upper limit)
3. Pregnant or breastfeeding, or positive pregnancy test in a pre-dose examination
4. Patients with known severe renal impairment (estimated glomerular filtration rate ≤30 mL/min/1.73 m2) or receiving continuous renal replacement therapy, hemodialysis, peritoneal dialysis
5. Will be transferred to another hospital which is not the study site within 72 hours.
6. Receipt of any experimental treatment for 2019-nCoV (off-label, compassionate use, or trial related) within the 30 days prior to the time of the screening evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
MTD | 28days(+/-2days)
  MTD is defined as highest dose level in which 6 subjects have been treated with less than 2 instances of DLT. DLT assessed during the study treatment period (28 ± 2 days) refers to a medically significant event which meets one of the criteria using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.

SECONDARY OUTCOMES:
Viral load | Time Frame: Day 1, 3, 5, 7, 9 and 12
  Viral load change (log10 viral load assessed by reverse transcription-qPCR)
Time to clinical improvement | Time Frame: dialy up to Day 10
  Assessed TTCI with WHO clinical progression scale by measuring clinical status daily. TTCI is defined as the time (in days) from initiation of study treatment until a decline of one category on WHO clinical progression scale which ranges from 0 (uninfected; no viral RNA detected) to 10 (death)

OTHER OUTCOMES:
Pharmacokinetic (PK) | Day 1,3 and 5.
  Cmax
Pharmacokinetic (PK) | Day 1,3 and 5.
  Ctrough
Pharmacokinetic (PK) | Day 1,3 and 5.
  AUCτ

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Seah, Study Director — J Ints Bio

IPD SHARING:
Plan to Share IPD: No